CLINICAL TRIAL: NCT00512044
Title: Local vs General Anaesthesia in Stapled Hemorrhoidectomy: A Multicentric Controlled Randomized Trial
Brief Title: Local Versus General Anaesthesia in Stapled Hemorrhoidectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment, internal problems with the study protocol
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, investigator, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07/CHV
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hemorrhoids
Keywords: anesthesia, Longo, mucosectomy, hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Anesthesia, Local; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: general (Active Comparator): general anesthesia: spinal and general
  Interventions: Procedure: general anesthesia (spinal and general)
- B: pudendal (Experimental): local anesthesia: pudendal block
  Interventions: Procedure: Local anesthesia (pudendal block)

INTERVENTIONS:
Procedure: Local anesthesia (pudendal block) — local anesthesia as indicated
  Other Names: local
  Arms: B: pudendal
Procedure: general anesthesia (spinal and general) — general according to guidelines
  Other Names: general
  Arms: A: general

SUMMARY:
The purpose of this study is to determine whether local or general anaesthesia in stapled hemorrhoidectomy leads to a shorter operation time with a better patient comfort.

DETAILED DESCRIPTION:
Hemorrhoids are a frequent disease with the need of surgical intervention in 10-20% of the patients. The stapled hemorrhoidectomy according to Longo under general anesthesia (or spinal) is considered standard of care [1]. Cohort studies show that a pudendal bloc with local anesthesia is safe and efficient [2-4]. The majority of procedures are actually performed in private clinics or in an ambulatory setting underlining the importance of economic issues such as procedure time (anesthesia and operation time) and hospital stay.

We hypothesize that stapled hemorrhoidectomy under local anaesthesia shortens anaesthesia time and hospital stay and reduces costs with no disadvantages regarding pain, satisfaction and complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Hemorrhoids grade III suitable for elective stapled hemorrhoidectomy

Exclusion Criteria:

* Age < 18 years
* No informed consent
* Emergency situation
* Contraindication to either anaesthesia method
* Patients not speaking french or german.
* Additional anal pathology (fissure, tumour).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Demartines, MD, Study Chair — Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland